CLINICAL TRIAL: NCT06115291
Title: Olfactory Training in Various Populations
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Jennifer Villwock, Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00146529
Record Dates: First submitted 2020-02-13; First posted 2023-11-02 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Olfactory Disorder; Smell Disorder; Traumatic Brain Injury; Concussion, Brain
MeSH Terms: conditions — Olfaction Disorders; Brain Injuries, Traumatic; Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: 4 scents (Experimental): Participants will be asked to inhale 4 different scents 2 times a day.
  Interventions: Other: Smell Test
- Group B: 14 scents (Active Comparator): Participants will be asked to inhale 14 different scents 2 times a day.
  Interventions: Other: Smell Test

INTERVENTIONS:
Other: Smell Test — Oils are used for each of the different scents. Each scent is administered via an aromatherapy inhaling stick.

SUMMARY:
To date, there is no validated pharmacotherapy for olfactory disorders. Interestingly, olfactory training - the intentional exposure to odorants for the purposes of retraining the sense of smell - has shown success with as many as 28% of subjects over the course of 12 weeks.

DETAILED DESCRIPTION:
Study Objectives: The overall, primary goals of these studies are as follows:

1. To compare the outcomes of our olfactory testing battery for olfactory training to the previously published literature
2. To determine if using a larger panel of odorants (our 15 scents versus the 4 scents previously used in the literature) yields a significant difference in olfactory recovery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Quantifiable or subjective olfactory dysfunction
* ability to complete objective olfactory tests and comply with olfactory training protocol

Exclusion Criteria:

* Anyone lower than the age of 18, or greater than the age of 80
* Pregnant women, as sinonasal symptoms and changes in smell can occur in pregnancy and are multifactorial
* Patients with poor or questionable compliance, as participation requires daily compliance with study protocol
* Patient's that are unable to perform routine follow-up
* Patients who are participating in another study during this trial
* Patients with dementia, Alzheimer's disease, Parkinson's disease, or other neurocognitive disorders, as these conditions are associated with baseline olfactory dysfunction.
* Patients with other systemic conditions known to impact the sinonasal cavity such as Wegener's granulomatosis, Churg Strauss, and immunodeficiency, as their impact on olfaction is unknown
* Patients who are allergic to any of the smells or components of our olfactory testing and training

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2020-02-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Olfactory Threshold | Change from baseline to month 6
  Changes in olfactory threshold when comparing pre- and post-olfactory training for performance in terms of percent correct per specific scent and overall combination of percent correct for all tested scents
Olfactory Identification | Change from baseline to month 6
  Changes in ability to detect and identify scents when comparing pre- and post-olfactory training for percent detected per individual scents and as a composite score reflecting performance on all scents

SECONDARY OUTCOMES:
Tolerance with Olfactory Training Protocol | At follow-up visits
  Self-reported tolerance with following olfactory training protocol
Neurocognition | Change from baseline to month 6
  Assessment of neurocognition and impact on olfactory quality of life using the Mini-Mental Status Exam (MMSE) and Montreal Cognitive Assessment (MoCA)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Villwock, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No